CLINICAL TRIAL: NCT04598074
Title: The Feasibility and Effectiveness of an Opioid Package Prototype (OPP) to Impact Opioid Prescribing, Dispensing, and Patient Use Outcomes
Brief Title: Opioid Package Prototype (OPP)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: University of Connecticut (Other); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nathaniel Rickles, Professor of Pharmacy Practice, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-210S-1; 75F40119C10152 (Other Grant/Funding Number: U.S. Food and Drug Administration)
Record Dates: First submitted 2020-10-07; First posted 2020-10-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use; Opioid Prescribing, Dispensing, and Patient Use
Keywords: oxycodone; opioid; opioids; package; packaging; post-surgical pain; post-operative pain; orthopedic; orthopaedic; surgery; dispensing; prescribing; blister; tablets; pain; opioid package prototype; OPP
MeSH Terms: conditions — Pain, Postoperative; Blister; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Package Prototype (OPP) (Experimental): Oxycodone 5mg tablets dispensed in the Opioid Package Prototype (OPP) with frequency and quantities varying, depending on the type of surgical procedure performed, surgeon, and individual patient
  Interventions: Other: Opioid Package Prototype (OPP)
- Usual Care (standard amber vial) (Active Comparator): Oxycodone 5mg tablets dispensed in the standard amber vial (usual care) with frequency and quantities varying, depending on the type of surgical procedure performed, surgeon, and individual patient
  Interventions: Other: Usual Care (standard amber vial)

INTERVENTIONS:
Other: Opioid Package Prototype (OPP) — The Opioid Package Prototype (OPP) is a child-resistant/senior-friendly, calendar-blister packaging of limited pill counts with flat readable billboard space for medication labeling.
  Arms: Opioid Package Prototype (OPP)
Other: Usual Care (standard amber vial) — The standard amber vial (orange bottle) is the container that medication is normally dispensed in outside of the study.
  Arms: Usual Care (standard amber vial)

SUMMARY:
The overall objective of this clinical trial is to identify the impact of selected package features, known as the Opioid Package Prototype (OPP), on the safe and effective use of opioids. Our specific aims are: (Aim 1) to evaluate the effectiveness of OPP on prescribing, dispensing, and patient use of oxycodone among orthopaedic surgery patients receiving post-operative outpatient oxycodone for post-surgical pain management, and (Aim 2) to determine the feasibility of OPP for orthopaedic surgery prescribers, pharmacists, and orthopaedic surgery patients. Such data can be used to further optimize packaging and labeling design, help patients and caregivers utilize their medication and packaging correctly, and improve prescribing and dispensing habits. The central hypothesis is that the OPP will be more effective than the amber vial in efforts to reduce oxycodone prescribing among patients over 18 receiving short-term management of post orthopedic surgery pain.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is 18 years and older;
2. The patient is one of the participating surgeons;
3. The patient is receiving orthopaedic surgery that involves the use of opioid medication for post-operative pain;
4. The patient is willing to receive oxycodone medication;
5. The patient is willing and able to receive medication at the UConn Health Specialty Pharmacy, located in the Exchange across the street from the main entrance of UConn Health;
6. The patient is willing and able to use a MyChart account;
7. The patient is able to read and understand English; and
8. The patient is able to understand the study procedures and their involvement in the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-09-07 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of tablets of oxycodone prescribed | 1 week after surgery
  Count via medical/pharmacy records
Number of tablets of oxycodone prescribed | 1 month after surgery
  Count via medical/pharmacy records
Number of tablets of oxycodone prescribed | 3 months after surgery
  Count via medical/pharmacy records
Average morphine milligram equivalent (MME) of oxycodone tablets prescribed/per participant | 1 week after surgery
  Mean
Average morphine milligram equivalent (MME) of oxycodone tablets prescribed/per participant | 1 month after surgery
  Mean
Average morphine milligram equivalent (MME) of oxycodone tablets prescribed/per participant | 3 months after surgery
  Mean
Number of oxycodone tablets used by study participants | 1 week after surgery
  Count via survey/interview/visual inspection/photograph
Number of oxycodone tablets used by study participants | 1 month after surgery
  Count via survey/interview/visual inspection/photograph
Number of oxycodone tablets used by study participants | 3 months after surgery
  Count via survey/interview/visual inspection/photograph
Average morphine milligram equivalent (MME) of oxycodone tablets used/per participant | 1 week after surgery
  Mean
Average morphine milligram equivalent (MME) of oxycodone tablets used/per participant | 1 month after surgery
  Mean
Average morphine milligram equivalent (MME) of oxycodone tablets used/per participant | 3 months after surgery
  Mean

SECONDARY OUTCOMES:
Number of requests for additional oxycodone prescriptions | 1 week, 1 month and 3 months after surgery
  Count per patient survey/interview
Amount of dispensing time per oxycodone prescription for each study participant | Time of surgery and any refills up to 1 month after surgery
  Log of dispensing start time (received prescription) and dispensing stop time (prescription ready for pick up)
Amount of counseling time per oxycodone prescription for each study participant | Time of surgery and any refills up to 1 month after surgery
  Log of counseling start time (start to discuss medication information) and counseling stop time (complete discussion of medication information)
Awareness of oxycodone tablets used | 1 week and 1 month after surgery
  Amount of time to report number of tablets used via brief inspection of container (not manual count) during interview and various survey questions
Change in knowledge of oxycodone from baseline to 1 week | Baseline (before surgery) and 1 week after surgery
  Number of correct answers out of 4 knowledge questions
Awareness of oxycodone medication information | 1 week and 1 month after surgery
  Various survey/interview questions
Consistency of access to oxycodone medication information | 1 week and 1 month after surgery
  Various survey/interview questions
SANE (Single Assessment Numeric Evaluation) score | Baseline, 1 week, 1 month and 3 months after surgery
  "How would you rate your affected joint/region of interest today as a percentage of normal (0% to 100% scale with 100% being normal)?"
PEG (Pain, Enjoyment of Life and General Activity) score | Baseline, 1 week, 1 month and 3 months after surgery
  A three-item scale assessing pain intensity and interference from 0-10. The three item scores are averaged for a final score and a higher number indicates greater pain and interference.
Pain Medication Attitudes Questionnaire (PMAQ-14) score | Baseline, 1 week, 1 month and 3 months after surgery
  Participants indicate the degree to which they agree with 14 statements regarding pain medication from 0 (never true) to 5 (always true). The 14 scores are averaged for a final score and a higher number indicates a more negative attitude toward pain medications,
Pain Catastrophizing Scale (PCS) | Baseline, 1 week, 1 month and 3 months after surgery
  A 13-item scale, with a total range of 0 to 52. Higher scores are associated with higher amounts of pain catastrophizing.
Peri-Operative Opioid-Related Symptom Distress Scale (OR-SDS) | 1 week, 1 month and 3 months after surgery
  A 4-point scale that evaluates 3 symptom distress dimensions (frequency, severity, bothersomeness) for 12 symptoms. The symptom-specific ORSDS is the average of the 3 symptom distress dimensions. The composite ORSDS is the average of 12 symptom-specific scores.
Patient Health Questionnaire-4 (PHQ-4) | Baseline, 1 week and 1 month after surgery
  A 4-item inventory rated on a 4-point Likert-type scale to assess for anxiety and depression. The minimum score (0) indicates no psychological distress and the maximum score (12) indicates severe psychological distress.
Feasibility of OPP for orthopaedic surgery prescribers | Within 1 month after prescribing the OPP to 30 participants
  Interview regarding benefits and weaknesses of the OPP design, interest in prescribing OPP in the future, and how OPP design can be improved for the future
Feasibility of OPP for pharmacists | After dispensing all OPPs (approximately 2 years)
  Interview questions regarding benefits and weaknesses of the OPP design, interest in dispensing OPP in the future, and how OPP design can be improved for the future
Feasibility of OPP for orthopaedic surgery patients | Between 1 and 3 months after surgery
  Interview questions regarding benefits and weaknesses of the OPP design, interest in using OPP in the future, and how OPP design can be improved for the future

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel M Rickles, PharmD, PhD, BCPP, FAPhA, Principal Investigator — University of Connecticut
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No